CLINICAL TRIAL: NCT07170670
Title: Cognitive-Behavioral Intervention Package for Port Catheter Needle Insertion: Effects on Pain, Anxiety, and Fear in Children With Cancer
Brief Title: Cognitive-Behavioral Care for Port Needle Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birgul Erdogan (Other)
Responsible Party: Sponsor-Investigator, Birgul Erdogan, Principal Investigator, Research Assistant, PhD, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024-25\04
Record Dates: First submitted 2025-08-19; First posted 2025-09-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cancer Associated Pain
Keywords: Pediatric Oncology; Port Catheter; Non-Pharmacological Intervention; Cognitive-Behavioral Intervention; Pain; Anxiety; Fear
MeSH Terms: conditions — Cancer Pain; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Intervention Package Group (Experimental): Before the procedure, children's pain, anxiety, and fear were assessed by the child, parent, and researcher. In the CBIP group, preparation, briefing, and implementation stages were conducted. The researcher met with the child and parent for preparation and briefing. A volunteer parent was trained to support the child during the procedure (e.g., sitting next to the child, holding hands, talking). Port catheter needle insertion was performed according to unit routine by the same nurse with 5 years' experience, using a single attempt. After the procedure, children rated pain (WB-FPRS), fear (CFS), and anxiety (CAS); the observing parent and researcher also completed CFS and CAS.
  Interventions: Behavioral: CBIP - Cognitive-Behavioral Intervention Package
- Control Group (No Intervention): In the study, children in the control group will receive the routine clinical procedure prior to the intervention, followed by port catheter needle insertion.

INTERVENTIONS:
Behavioral: CBIP - Cognitive-Behavioral Intervention Package — Before the procedure, the researcher initiated social interaction with the child (cognitive distraction). Next, suggestions regarding the procedure were provided (guidance). A volunteer parent sat beside the child, providing support by holding the child's non-procedural hand. While the nurse performed the port catheter insertion, the researcher applied one of the behavioral distraction techniques chosen by the child during the pre-procedure phase, such as counting, singing, reading a poem, or answering questions (behavioral distraction). Upon completion of the procedure, the researcher provided positive reinforcement by praising the child ("Well done!" and "You were very brave!") and rewarding the child with a star and smiley face sticker on the collar (positive reinforcement).
  Arms: Cognitive-Behavioral Intervention Package Group

SUMMARY:
This study aims to determine the effect of the Cognitive-Behavioral Intervention Package (CBIP) applied during port catheter needle insertion on pain, anxiety, and fear levels in children aged 6-18 years diagnosed with oncology.

Research Hypotheses

Between the Cognitive-Behavioral Intervention Package group (G1) and the control group (G2):

H1: There is a difference in the mean scores of the Wong-Baker FACES Pain Rating Scale (WB-FPRS) between the groups.

H2: There is a difference in the mean scores of the Children's Anxiety Scale between the groups.

H3: There is a difference in the mean scores of the Children's Fear Scale between the groups.

Prior to the intervention, researchers will administer the scales to the intervention group, followed by the implementation of the CBIP. After the port catheter needle insertion, the scales will be re-administered to evaluate the final levels of pain, anxiety, and fear.

ELIGIBILITY:
Inclusion Criteria:

* Are 6-18 years old,
* Have a cancer diagnosis,
* Have undergone at least one prior port catheter needle insertion,
* Are willing to participate along with parental consent.

Exclusion Criteria:

* Have any visual, auditory, verbal, or cognitive impairment,
* Are in the terminal stage of the disease,
* Have a history of sedative, analgesic, or narcotic use within 24 hours prior to enrollment,
* Have a fever or history of infection at the time of enrollment,
* Have a pre-procedure WB-FPRS score of 2 or higher unrelated to the procedure,
* Do not complete the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Characteristics Form (SCF) | At baseline, prior to intervention (Day 1)
  The form was developed by the researchers based on the literature. It consists of 11 questions addressing the sociodemographic characteristics of parents and children, as well as the status of port catheter needle insertion.
Wong-Baker FACES Pain Rating Scale (WB-FPRS) | Before and after port catheter needle insertion (Day 1).
  Pain will be assessed using the Wong-Baker FACES Pain Rating Scale (WB-FPRS) and completed by the child before and after the port catheter needle insertion. Scores range from 0 to 5, where 0 indicates no pain and 5 indicates unbearable pain.
Children's Fear Scale (CFS) | Before and after port catheter needle insertion (Day 1).
  Fear will be assessed using the Children's Fear Scale (CFS) by the child, parent, and researcher before and after the port catheter needle insertion. Scores range from 0 to 4, where 0 indicates no fear and 4 indicates extreme fear.
Children's Anxiety Scale-State (CAS-S) | Before and after port catheter needle insertion (Day 1).
  Anxiety will be assessed using the Children's Anxiety Scale-State (CAS-S) as reported by the child, parent, and researcher before and after the port catheter needle insertion. Scores range from 0 to 5, where 0 indicates no anxiety and 5 indicates extreme anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Faculty of Health Sciences, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No